CLINICAL TRIAL: NCT04720404
Title: Mindful Prevention of Psychopathology in Healthcare Workers During the COVID-19 Crisis (COVID-19 MindPreP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Anne Speckens, Professor Anne Speckens, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MFN-COVID-19 2020-22
Record Dates: First submitted 2021-01-12; First posted 2021-01-22 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Mindfulness; Randomized Controlled Trial; Psychopathology; Health Personnel
Keywords: COVID-19; Mindfulness-Based Stress Reduction; Healthcare workers; Positive Mental Health; Working mechanisms
MeSH Terms: conditions — COVID-19 | interventions — Mindfulness-Based Stress Reduction; Palliative Care

STUDY DESIGN:
Intervention Model Description: Randomized, controlled clinical trial of interactive MBSR program added to support as usual (MBSR + SAU) versus support as usual with daily self-help mindfulness exercises via a YouTube-channel (SAU + DMYT)
Who Masked: Outcomes Assessor
Masking Description: Outcomes on psychiatric interview will be assessed by independent research assistants blind to condition. Participants will be instructed to avoid unblinding as much as possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction program (Experimental): Healthcare workers in the MBSR arm will be invited to participate in an adapted online MBSR program added to support as usual
  Interventions: Behavioral: Mindfulness-Based Stress Reduction; Other: Support as usual
- Daily self-help mindfulness exercises via YouTube-channel (Active Comparator): Healthcare workers in the self-help arm will be invited to follow a self-help program with mindfulness/compassion exercises of 30 minutes per day via YouTube channel
  Interventions: Other: Self-help mindfulness/compassion exercises; Other: Support as usual

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — Participants in the intervention group will follow a 4-week adapted MBSR training. The training consists of biweekly sessions of 1,5 hours. The training is structured based on the Mindfulness-Based Stress Reduction training as originally designed by John Kabat Zinn. The program includes both formal and informal meditation exercises.
  Other Names: MBSR; Mindfulness-based Intervention
  Arms: Mindfulness Based Stress Reduction program
Other: Self-help mindfulness/compassion exercises — Participants in the self-help group will receive a 4-week program with daily suggestions for mindfulness/compassion exercises of 30 minutes on a YouTube-channel. Participants can schedule the exercises themselves.
  Arms: Daily self-help mindfulness exercises via YouTube-channel
Other: Support as usual — Support as usual (SAU) consists of facilities or interventions already available healthcare organisations provided to their healthcare workers (e.g. buddy-, team- and peer support system, shopping/dinner service etc.).

SUMMARY:
The current study will be a randomized controlled trial (RCT) investigating an adapted online Mindfulness-Based Stress Reduction (MBSR) program versus daily online self-help mindfulness exercises, in preventing incident/prevalent psychopathology in healthcare workers allocated to work with COVID-19 patients. Outcome measures include depression, anxiety, somatoform symptoms, post-traumatic stress, insomnia, substance abuse, post-traumatic growth and positive mental health. The study also aims to explore possible working mechanisms such as perseverative thinking, mindfulness skills and self-compassion.

The study will have a follow-up duration of 7 months from baseline.

DETAILED DESCRIPTION:
Introduction With the rapid developments to anticipate and manage the ongoing COVID-19 pandemic, healthcare personnel is quickly reallocated to COVID-19 units. These people will experience substantial amounts of stress which has been shown to result in the development or increase of stress related disorders like psychological distress and psychopathology in 50-70%. Adaptive reconsolidation of stressful events is required for resilience against prolonged stress and prevent development and/or recurrence of psychopathology.

Mindfulness-based interventions (MBIs) are potent interventions with profitable results in many people with and without stress-related disorders. These interventions invite people to allow bodily sensations, thoughts and feelings in reaction to and in the aftermath of stressors and pay attention to them in a particular way: on purpose, in the present moment, and without judgment. The effectiveness of these interventions on stress reduction is now founded on a strong meta-analytical evidence base in symptom and stress-reduction in diverse clinical and non-clinical populations.

Mindfulness-based Stress Reduction (MBSR) is a specific stress-focused MBI. In healthcare professionals, MBSR training increased well-being, mindfulness skills, empathy and emotional stability and decreased burnout, anxiety, and depression. A randomized clinical trial showed that specifically residents with high baseline levels of emotional exhaustion benefitted from MBSR. Moreover, MBSR can be delivered effectively via interactive video-conferencing, which makes it suited to quickly support relatively large groups of healthcare workers.

Taken together that MBSR has beneficial effects in healthcare workers and is aimed at dealing with stress, this makes it a potentially useful intervention to prevent psychopathological sequela of the high-stress situations for healthcare workers inherent to the current COVID-19 outbreak. However, the effectiveness of an additional MBSR intervention in a severe crisis situation like the COVID-19 outbreak needs to be empirically investigated in a prospective study, before large scale implementation is advocated.

Aims The aim of the study is to investigate the effectiveness of an adapted online MBSR added to Support As Usual (SAU) versus daily self-help mindfulness exercises via a YouTube-channel (DMYT) + SAU on the incidence and prevalence of psychological distress and psychopathology (anxiety, depression, somatoform symptoms). In addition, we aim to decrease post-traumatic stress symptoms, insomnia, substance abuse and health-related costs more in the MBSR + SAU group. We also aim to improve the post-traumatic growth, positive mental health and health-related quality of life. Furthermore, we will investigate whether improving mindfulness skills and self-compassion and decreasing repetitive negative thinking may help reduce psychological distress (working mechanism).

Method A two-armed randomized, controlled superiority trial comparing an adapted MBSR + SAU versus DMYT + SAU for reducing psychological distress and psychopathology in healthcare workers working with COVID-19 patients. Assessments will be conducted at baseline, post intervention (1 month) and follow-up at 4 and 7 months.

The intervention is an interactive adapted online MBSR program. The training consists of eight 1.5 hour group sessions twice per week during 4 weeks and daily home practice assignments guided by audio files. The sessions will be held via interactive video-streaming. MBSR courses will be taught by qualified mindfulness teachers. Participants in the control condition will have the possibility to use a self-help daily mindfulness exercise of 30 minutes on a YouTube channel (DMYT) for 4 weeks. Both will be offered on top of the other interventions (SAU) already available in the hospital or organization (e.g. buddy-, team- and peer support system, shopping/dinner service, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers who are either currently or in past have been working directly with COVID-19 patients, e.g. on COVID-19 ward/intensive care unit.

Exclusion Criteria:

* Impossibility to obtain a valid informed consent
* Insufficient comprehension of the Dutch language
* Inability to access the interactive videoconferencing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Somatoform symptoms, Anxiety, Depression | Change between baseline and 7 months
  Measured by the Patient Health Questionnaire - Somatoform symptoms, Anxiety, Depression (PHQ-SADS). The PHQ-SADS is a 31-item self-reported measure combining 3 questionnaires, the 9-item Patient Health Questionnaire (PHQ-9), the 7-item Generalized Anxiety Disorder scale (GAD-7) and the 15-item Patient Health Questionnaire (PHQ-15). The PHQ-9 is designed to measure depression in general medical and mental health settings. The GAD-7 measures severity of anxiety. The PHQ-15 is used to screen for somatization and monitoring somatic symptoms severity.

SECONDARY OUTCOMES:
Occurence of psychopathology | At 7-months follow-up
  This will be assessed by a Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-V). This diagnostic instrument assess occurence of depression, anxiety disorder, PTSS, substance abuse and somatoform disorder.
Post-traumatic stress symptoms | At baseline, 1, 4 and 7 months
  Measured by the PTSS Checklist for the DSM-5 (PCL-5). This is a 20-item self-report measure to assess the 20 DSM-5 symptoms of post-traumatic stress disorder.
Severity of insomnia | At baseline, 1, 4 and 7 months
  Measured by the Insomnia Severity Index (ISI), a 7-item self-reported screening measure for insomnia.
Alcohol use | At baseline, 1, 4 and 7 months
  Measured by the Alcohol Use Disorders Identification Test (AUDIT-C) consisting of 10 items being a screening method for unhealthy alcohol use.
Posttraumatic growth | At baseline, 1, 4 and 7 months
  Measured by the Posttraumatic Growth Inventory-Short Form (PTGI-SF). The PTGI-SF is a 10-item questionnaire and measures the general tendency to experience difficult events in such a way that benefits are perceived.
Positive mental health | At baseline, 1, 4 and 7 months
  Measured by the Mental Health Continuum-Short Form (MHC-SF). The MHC-SF is a questionnaire consisting of 14 items measuring emotional, social and psychological well-being.
Health-related quality of life | At baseline, 1, 4 and 7 months
  Measured by the EuroQol-5D-5L. The EQ-5D-5L consist of five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems and extreme problems).
Costs | At 7 months follow-up
  This will be investigated by using the Treatment Inventory Costs associated with Psychiatric Illness (TiC-P) as a measure of healthcare utilization.

OTHER OUTCOMES:
Mindfulness skills | At baseline, 2 weeks, 1, 4 and 7 months
  Measured by the 24-item Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) divided into the subscales observing, describing, acting with awareness, non-judging and non-reactivity.
Self-compassion | At baseline, 2 weeks, 1, 4 and 7 months
  Measured by the 12-item Dutch Self-Compassion Scale - Short Form (SCS-SF) consisting of six components, including self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification.
Repetitive negative thinking | At baseline, 2 weeks, 1, 4 and 7 months
  Measured by the 15-item Perseverative Thinking Questionnaire (PTQ)PTQ consists of 15-items and assess repetitive negative thinking.
Mindfulness practice | At baseline, 2 weeks, 1, 4 and 7 months
  This questionnaire lists the intensity and form of formal and informal mindfulness exercises the participant conducted in the past 2 months at baseline, or in-between the questionnaires for the other follow-up measures. In addition, this list makes an inventory of whether participants have followed another intervention in addition to the mindfulness intervention offered in this study.
Covid-related aspects | At baseline, 1, 4 and 7 months
  A variety of facets related to COVID-19 (work, society and person-related) will be elucidated by a 21-item questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Speckens, Prof., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The authors intend to make the data available to other researchers after completion of the study and will comply with open access procedures, including open access publishing as much as possible.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: We expect the final report of the primary endpoint of the study in May 2022, and we will have an embargo period of 6 months after publication.
Access Criteria: We will use restricted access, such that interested researchers are welcome to contact us with requests for data. The project team will review the quality of the request and grant permission if the request is in accordance with the terms of use drafted by the Radboudumc.
URL: http://www.lcrdm.nl

REFERENCES:
- [Background] Bohlmeijer E, ten Klooster PM, Fledderus M, Veehof M, Baer R. Psychometric properties of the five facet mindfulness questionnaire in depressed adults and development of a short form. Assessment. 2011 Sep;18(3):308-20. doi: 10.1177/1073191111408231. Epub 2011 May 17. PMID 21586480
- [Background] Cann A, Calhoun LG, Tedeschi RG, Taku K, Vishnevsky T, Triplett KN, Danhauer SC. A short form of the Posttraumatic Growth Inventory. Anxiety Stress Coping. 2010;23(2):127-37. doi: 10.1080/10615800903094273. PMID 19582640
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. The Patient Health Questionnaire Somatic, Anxiety, and Depressive Symptom Scales: a systematic review. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):345-59. doi: 10.1016/j.genhosppsych.2010.03.006. Epub 2010 May 7. PMID 20633738
- [Background] Lamers SM, Westerhof GJ, Bohlmeijer ET, ten Klooster PM, Keyes CL. Evaluating the psychometric properties of the Mental Health Continuum-Short Form (MHC-SF). J Clin Psychol. 2011 Jan;67(1):99-110. doi: 10.1002/jclp.20741. PMID 20973032
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Schippers GM, Broekman TG, Buchholz A, Koeter MW, van den Brink W. Measurements in the Addictions for Triage and Evaluation (MATE): an instrument based on the World Health Organization family of international classifications. Addiction. 2010 May;105(5):862-71. doi: 10.1111/j.1360-0443.2009.02889.x. Epub 2010 Mar 10. PMID 20331557
- [Background] Weathers, F.W., Litz, B.T., Keane, T.M., Palmieri, P.A., Marx, B.P., & Schnurr, P.P. (2013). The PTSD Checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD at www.ptsd.va.gov.
- [Background] Ehring T, Zetsche U, Weidacker K, Wahl K, Schonfeld S, Ehlers A. The Perseverative Thinking Questionnaire (PTQ): validation of a content-independent measure of repetitive negative thinking. J Behav Ther Exp Psychiatry. 2011 Jun;42(2):225-32. doi: 10.1016/j.jbtep.2010.12.003. Epub 2010 Dec 21. PMID 21315886
- [Background] Lai J, Ma S, Wang Y, Cai Z, Hu J, Wei N, Wu J, Du H, Chen T, Li R, Tan H, Kang L, Yao L, Huang M, Wang H, Wang G, Liu Z, Hu S. Factors Associated With Mental Health Outcomes Among Health Care Workers Exposed to Coronavirus Disease 2019. JAMA Netw Open. 2020 Mar 2;3(3):e203976. doi: 10.1001/jamanetworkopen.2020.3976. PMID 32202646
- [Background] Goldberg SB, Tucker RP, Greene PA, Davidson RJ, Wampold BE, Kearney DJ, Simpson TL. Mindfulness-based interventions for psychiatric disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2018 Feb;59:52-60. doi: 10.1016/j.cpr.2017.10.011. Epub 2017 Nov 8. PMID 29126747
- [Background] Khoury B, Sharma M, Rush SE, Fournier C. Mindfulness-based stress reduction for healthy individuals: A meta-analysis. J Psychosom Res. 2015 Jun;78(6):519-28. doi: 10.1016/j.jpsychores.2015.03.009. Epub 2015 Mar 20. PMID 25818837
- [Background] Krasner MS, Epstein RM, Beckman H, Suchman AL, Chapman B, Mooney CJ, Quill TE. Association of an educational program in mindful communication with burnout, empathy, and attitudes among primary care physicians. JAMA. 2009 Sep 23;302(12):1284-93. doi: 10.1001/jama.2009.1384. PMID 19773563
- [Background] Shapiro SL, Schwartz GE, Bonner G. Effects of mindfulness-based stress reduction on medical and premedical students. J Behav Med. 1998 Dec;21(6):581-99. doi: 10.1023/a:1018700829825. PMID 9891256
- [Background] Verweij H, van Ravesteijn H, van Hooff MLM, Lagro-Janssen ALM, Speckens AEM. Mindfulness-Based Stress Reduction for Residents: A Randomized Controlled Trial. J Gen Intern Med. 2018 Apr;33(4):429-436. doi: 10.1007/s11606-017-4249-x. Epub 2017 Dec 18. PMID 29256091
- [Background] Kabat-Zinn J, Full Catastrophe Living (Revised Edition): Using the wisdom of your body and mind to face stress, pain, and illness. 2013. Random House Publishing Group.
- [Derived] Arts-de Jong M, Geurts DEM, Spinhoven P, Ruhe HG, Speckens AEM. Mindfulness-Based Interventions for Mental Health Outcomes in Frontline Healthcare Workers During the COVID-19 Pandemic: A Randomized Controlled Trial. J Gen Intern Med. 2025 Nov;40(15):3705-3714. doi: 10.1007/s11606-025-09529-z. Epub 2025 May 19. PMID 40388083

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT04720404/SAP_000.pdf